CLINICAL TRIAL: NCT01487577
Title: A Pilot Study of Pharmacokinetics-based Mycophenolate Mofetil Dosing for Graft-Versus-Host-Disease Prophylaxis in Pediatric Blood and Marrow Transplantation
Brief Title: Pharmacokinetics-based Mycophenolate Mofetil Dosing for GVHD Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Randy Windreich, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHP_BMT_MMF_10
Record Dates: First submitted 2011-11-23; First posted 2011-12-07 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Allogeneic Blood and Marrow Transplantation (BMT); Graft Versus Host Disease
Keywords: Allogeneic blood and marrow transplantation (BMT); Graft versus host disease; Mycophenolate mofetil; Pharmacokinetics
MeSH Terms: conditions — Graft vs Host Disease | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mycophenolate mofetil (Experimental): Pharmacokinetics-based targeting of mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — Based on individual pharmacokinetics data, mycophenolate mofetil will be administered by continuous infusion to target a desired AUC exposure
  Other Names: Cellcept; MMF

SUMMARY:
Bone marrow transplantation (BMT) is used to successfully treat high-risk forms of leukemia, lymphoma, and other childhood cancers that were once considered incurable. A major barrier to the application of this life-saving treatment is acute graft-versus-host disease (GVHD) which develops in approximately 30-80% of patients and is a leading cause of death from transplant complications. Current GVHD prevention methods are not very efficacious and lead to unacceptable side effects. Mycophenolate mofetil (MMF), an anti-rejection medication used in solid organ transplants, has shown great promise in BMT recipients. The effectiveness of MMF depends on blood levels of mycophenolic acid (MPA, the active form of MMF). Different patients have been found to have different blood levels of MPA when they are given the same dose of MMF. The purpose of this study is to study a novel method of giving MMF based on its metabolism (pharmacokinetics) to achieve desired blood levels of MPA for prevention of GVHD. Non-invasive ways of monitoring the drug exposure will also be studied. The ultimate goal of this study is to improve approaches to GVHD prevention and improve outcomes of BMT in children.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) remains a major barrier to the success of allogeneic blood and marrow transplant (BMT) therapy. Acute GVHD is seen in 30-80% of patients and once established, often responds poorly to therapy and is associated with chronic disease and increased risk of death. Although combination of methotrexate (MTX) and a calcineurin inhibitor has been the "standard of care" for more than a quarter of a century, there is little consensus on the most effective and least toxic approach to GVHD prevention. MTX use is associated with painful mucositis, delay in engraftment and potential pulmonary toxicity. For cord blood transplants, commonly, a calcineurin inhibitor is used with corticosteroids and antithymocyte globulin. Steroid therapy is frequently complicated by high rates of infection, hyperglycemia and hypertension.

Mycophenolate mofetil (MMF), whose metabolite mycophenolic acid (MPA) inhibits proliferation of lymphocytes, is approved for prevention of organ transplant rejection. MMF in combination with CsA is widely used for GVHD prevention in patients receiving reduced-intensity conditioning BMT. It has also been successfully used in primary and salvage therapy of acute GVHD. In myeloablative transplants, while the GVHD outcomes appear comparable, this regimen appears to have superior toxicity profile in comparison to CsA and MTX with faster hematopoietic engraftment and reduced severity and duration of mucositis.

One challenge with MMF use in BMT recipients is a significantly lower MPA exposure in the immediate post-conditioning period when compared to organ transplant recipients. This has been shown in a number of pharmacokinetics studies including our preliminary data on pediatric myeloablative transplants. Low total and unbound MPA trough concentrations are associated with higher rates of acute GVHD and graft rejection, and lower response rates in treatment of acute GVHD. There is also poor correlation between MPA trough concentration and area under the concentration curve (AUC). While most previous studies have used fixed MMF dosing, one recent study in adults has shown feasibility of AUC-based individualized MMF dosing.

This protocol is based on the premise that optimization of MPA exposure in the immediate post-transplant phase will lead to better acute GVHD prevention. It will study an AUC-based targeting of MMF in pediatric patients undergoing myeloablative allogeneic BMT. We propose a novel continuous infusion method for MMF administration to achieve total MPA steady state concentration. Salient findings emerging from this study will be examined and in replicate cohorts of pediatric and adult patients undergoing allo-BMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 6 months and 21 years of age.
* Recipients of an allogeneic blood and marrow transplant (BMT).
* Stem cell sources should be bone marrow or umbilical cord blood.
* Bone marrow or cord blood unit: Sibling should be HLA matched at A, B and DRB1 loci. Unrelated cord blood unit should be at a minimum 4/6 matched at allele level on HLA A, B and DRB1 loci. Unrelated donor should be HLA allele level matched at A, B, C and DRB1 loci.
* Minimum prefreezing nucleated cell dose for cord blood units: 3x10^7/kg for malignant diseases and 5x10^7/kg for nonmalignant diseases.
* Conditioning regimen must be myeloablative in intensity. Examples include but are not limited to Cy/TBI, BuCy 200, etc.
* Patients ≥ 16 years old must have a Karnofsky score ≥ 70%, and patients < 16 years old must have a Lansky score ≥ 70%.
* Renal: Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2.
* Hepatic: Total bilirubin ≤ 2.5 mg/dL unless the increase in bilirubin is attributable to Gilbert's syndrome; and SGOT (AST), SGPT (ALT), and Alkaline Phosphatase < 5 x upper limit of normal (ULN) for age.
* Cardiac: Left ventricular ejection fraction at rest > 40%, or shortening fraction > 26%, by echocardiogram or radionuclide scan.
* Pulmonary: FEV1, FVC, and DLCO (diffusion capacity) > 50% of predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation > 92% of room air.

Exclusion Criteria:

* Patients with a known hypersensitivity to MMF.
* Prior autologous or allogeneic BMT < 12 months prior to enrollment.
* Mismatched related donor.
* Mismatched unrelated marrow donor.
* Peripheral blood stem cell source.
* Reduced intensity conditioning.
* Uncontrolled bacterial, viral, fungal or other infection.
* Evidence of HIV infection or HIV positive serology.
* Requirement of supplemental oxygen.
* Patients who are pregnant (B-hCG positive) or breastfeeding. All females of 11 years of age or older and/or who have begun menstruating will be screened for hCG by either urinalysis or a blood sample in order to screen for pregnancy status, as per institutional BMT policy.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy M Windreich, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Candidates are identified through the investigators' clinical practice.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil
Started | 19
Completed | 18 (One participant became ineligible after signing consent, but before receiving protocol therapy.)
Not Completed | 1
Not completed — Became ineligible after signing consent | 1

BASELINE CHARACTERISTICS:
Population: Pediatric hematopoietic stem cell recipients undergoing myeloablative conditioning therapy
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade ≥3 Toxicities Scored According to the CTCAE Version 4.0.
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants | 0

2. Primary Outcome: Number of Participants With Acute Grade II-IV GVHD, Acute Grade III-IV GVHD, and Chronic GVHD.
Description: Acute GVHD will be graded according to the Modified Glucksberg Staging Criteria. Chronic GVHD will be graded according to NIH Chronic GVHD Consensus Guidelines.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants
  Acute grade II-IV GVHD | 6
  Acute grade III-IV GVHD | 4
  Chronic GVHD | 2

3. Secondary Outcome: Number of Participants With Neutrophil and Platelet Engraftment.
Description: Neutrophil and platelet engraftment definitions as defined by the CIBMTR Data Management Manual.
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants
  Incidence of neutrophil engraftment | 18
  Incidence of platelet engraftment | 15

4. Secondary Outcome: Number of Participants Who Experienced Relapse.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants | 4

5. Secondary Outcome: Number of Participants Who Experienced Nonrelapse Mortality.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants | 0

6. Secondary Outcome: Number of Participants in Overall Survival.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
participants | 15

7. Secondary Outcome: Pharmacokinetic Analysis of MMF AUC to Evaluate MMF Dose Relationships to Drug Exposure.
Description: Pharmacokinetic analysis includes, but is not limited to, area under the plasma concentration versus time curve (AUC).
Time Frame: 100 days
Measure: Median (Full Range); unit: mcg*hr/mL
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
mcg*hr/mL
  AUC, Intermittent IV dosing | 46.5 [16.7 to 65.9]
  AUC, Continuous infusion | 40.1 [20.6 to 63.8]
  AUC, Intermittent PO dosing | 36.1 [11.9 to 95.9]

8. Secondary Outcome: Pharmacokinetic Analysis of MMF Clearance to Evaluate MMF Dose Relationships to Drug Exposure.
Description: Pharmacokinetic analysis includes, but is not limited to, clearance.
Time Frame: 100 days
Measure: Median (Full Range); unit: mL/min/kg
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
mL/min/kg
  Clearance, Intermittent IV dosing | 10.2 [6.8 to 30.8]
  Clearance, Continuous infusion | 15.1 [7.2 to 73]
  Clearance, Intermittent PO dosing | 10.9 [4.9 to 26.6]

9. Secondary Outcome: Pharmacokinetic Analysis of MMF Steady State Concentration to Evaluate MMF Dose Relationships to Drug Exposure.
Description: Pharmacokinetic analysis includes, but is not limited to, steady-state concentrations.
Time Frame: 100 days
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 18
mcg/mL
  Steady-state concentration, Intermittent IV dosing | 1.9 [0.6 to 2.7]
  Steady-state concentration, Continuous infusion | 1.7 [0.9 to 2.7]
  Steady-state concentration, Intermittent PO dosing | 1.5 [0.5 to 4.0]

ADVERSE EVENTS:
Time Frame: 1 year post-enrollment
Arm/Group | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (N=18)
Tracheitis (Infections and infestations) | 1 (1) — Laryngotracheitis due to HSV
Hepatobiliary disorders, other (Hepatobiliary disorders) | 2 (2) — Veno-occlusive disease of the liver
Pericardial effusion (Cardiac disorders) | 1 (1) — Aseptic pericardial effusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (N=18)
Acute GVHD (Immune system disorders) | 8 (8)
Chronic GVHD (Immune system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Our study is limited by small sample size and heterogeneity in stem cell sources. Besides targeted MMF dosing, other factors that might have affected clinical outcomes include duration of MMF and use of ATG in unrelated-donor transplants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes